CLINICAL TRIAL: NCT01509885
Title: Phase 3 Study of Cyproheptadine and Chlorpromazine Effects on Spasticity After Spinal Cord Injury
Brief Title: Cyproheptadine and Chlorpromazine Effects on Spasticity
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00020682
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Spinal Cord Injuries; Muscle Spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

GROUPS / COHORTS (2):
- Complete Spinal Cord Injured Subjects: Patients with no motor scores in their legs and suffering a complete spinal cord injury.
- Incomplete Spinal Cord Injured Subjects: Patient with some motor preservation below the injury and suffering an incomplete spinal cord injury.

SUMMARY:
The main goal of this research is to understand the neuronal mechanisms that mediate the development of spasticity and motor dysfunction after spinal cord injury. The investigators examine how neurons and neuronal circuits in an injured nervous system adapt to produce the uncontrolled and unwanted muscle contractions that affect the majority (80%) of patients with spinal cord injury. One of the neurons that the investigators study is the motoneuron that excites the muscles of the limbs to produce movement. Previously, the investigators have shown that after spinal cord injury, the excessive and uncontrolled activity of motoneurons during muscle spasms is mediated, in large part, by the activation of calcium currents in the human motoneuron. In human patients the investigators have used recordings from single muscle fibres to estimate the contribution of these calcium currents in activating the motoneuron during muscle spasms. In this proposal, the investigators study why motoneurons recover these calcium currents and self-sustained activity after chronic spinal cord injury. Because the calcium currents require the presence of the monoamine serotonin (5HT) to activate, and this monoamine is greatly reduced after injury, the investigators examine if the calcium currents recover because the 5HT receptors become spontaneously active without the need for 5HT to bind to the receptor, which the investigators hypothesize to be one of the causes of spasticity after spinal cord injury. This research will pave the way to develop new pharmacological and rehabilitative therapies to both control spasticity after spinal cord injury and augment residual motor movements.

ELIGIBILITY:
Inclusion Criteria:

Patients must have suffered a trauma to the spinal cord at least 6 months ago or longer. In addition, subjects must exhibit some degree of spasticity as determined by having an Ashworth Spasticity Score, as assessed by a physical therapist, greater than 1.

Exclusion Criteria:

* If patients have damage to the nervous system other than to the spinal cord
* Pregnant women
* Elderly Patients and debilitated patients
* Alcoholic Patients
* Patients with:

  * Known or suspected allergy to the medication or its ingredients
  * Cardiovascular disease
  * Hypotension
  * Coronary artery disease
  * Reduced liver or kidney function
  * Comatose or depressed states due to CNS depressants
  * Blood dyscrasias
  * Bone marrow depression
  * History of seizures
  * Respiratory problems
  * Hypocalcemia
  * Monoamine oxidase inhibitor therapy
  * Angle-closure glaucoma
  * Stenosing peptic ulcer
  * Symptomatic prostatic hypertrophy
  * Bladder neck obstruction
  * Pyloroduodenal obstruction
  * History of bronchial asthma
  * Increased intraocular pressure
  * Hyperthyroidism
  * Cardiovascular disease
  * Hypertension
* Patients taking:

  * Amphetamines
  * Antihistamines-second generation
  * Anticonvulsants
  * Anticholinergics
  * CNS depressants
  * Antidepressants
  * Hypotensive agents
  * Levodopa
  * Lithium

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Spinal Cord Injury Patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cutaneomuscular Reflex Responses | Change after drug intake at baseline, 30minutes, 60minutes, 90minutes and 120minutes
  Tibialis anterior reflex responses evoked by stimulation of the medial arch of the foot will be measured before and after drug administration.
Paired motor unit recordings | Change at baseline and 30, 60, 90 and 120min after drug intake
  We obtain paired motor unit recordings to determine changes in neuronal excitability after drug intake in incomplete spinal-cord injured subjects only.

SECONDARY OUTCOMES:
Blood pressure and Heart rate | Change at baseline and 30, 60, 90, 120 minutes after drug intake
  We measure blood pressure and heart rate to determine the safety of the drug during the experiment and whether we can continue safely.

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Gorassini, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Murray KC, Nakae A, Stephens MJ, Rank M, D'Amico J, Harvey PJ, Li X, Harris RL, Ballou EW, Anelli R, Heckman CJ, Mashimo T, Vavrek R, Sanelli L, Gorassini MA, Bennett DJ, Fouad K. Recovery of motoneuron and locomotor function after spinal cord injury depends on constitutive activity in 5-HT2C receptors. Nat Med. 2010 Jun;16(6):694-700. doi: 10.1038/nm.2160. Epub 2010 May 30. PMID 20512126
- See also: Related Info — http://www.scialberta.ca/